CLINICAL TRIAL: NCT06024252
Title: Efficacy, Safety, and Treatment Patterns of Transcatheter Arterial Chemoembolization (TACE) Combined With Atezolizumab and Bevacizumab in Unresectable Hepatocellular Carcinoma: a Multicenter, Retrospective, Observational Real-world Study
Acronym: CHANCE023
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dr. Gao-Jun Teng, Zhongda Hospital
Other Study IDs: CHANCE023
Record Dates: First submitted 2023-08-06; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: HCC
MeSH Terms: interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: TACE — TACE in combination with atezolizumab + bevacizumab for at least one interval of no more than eight weeks.
  Other Names: Atezolizumab; Bevacizumab

SUMMARY:
This study will evaluate the efficacy and safety of TACE combined with atezolizumab + bevacizumab in the treatment of unresectable hepatocellular carcinoma, and the treatment patterns of the combination regimen

DETAILED DESCRIPTION:
This study is a multi-center, retrospective and observational real-world study to explore the efficacy, safety and treatment pattern of TACE combined with Atezolizumab + Bevacizumab in unresectable hepatocellular carcinoma. The target population for the planned retrospective analysis of this project is patients who have been diagnosed with unresectable HCC according to the guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2019 Edition) and treated with TACE combined with atezolizumab + bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. All patients were diagnosed with unresectable hepatocellular carcinoma according to the guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2019 Edition);
2. Patients ≥ 18 years old, male or female;
3. Child-Pugh Class A and B liver function;
4. ECOG-PS score of 0 ~ 2 points;
5. Received TACE in combination with atezolizumab + bevacizumab for at least one interval of no more than eight weeks.

Exclusion Criteria:

1. Other primary malignancies;
2. Incomplete data, such as no baseline image that can be assessed according to RECIST 1.1 or mRECIST, and survival outcome.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population for the planned retrospective analysis of this project is patients who have been diagnosed with unresectable HCC according to the guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2019 Edition) and treated with TACE combined with atezolizumab + bevacizumab.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Overall survival (OS): defined as the time from the start of the first TACE or atezolizumab + bevacizumab (whichever occurs first) to death due to any cause.

SECONDARY OUTCOMES:
Progression-Free Survival | 1 year
  Progression-Free Survival (PFS): defined as the time from the start of the first TACE or atezolizumab + bevacizumab (whichever occurs first) to the first occurrence of disease progression or death from any cause.
Objective response rate | 1 year
  Objective response rate (ORR): defined as the percentage of patients with objective response (CR and PR) from the start of treatment until tumor progression.
One-year survival rate | 1 year
  One-year survival rate: defined as the percentage of patients who are survival for 1 year from the start of this treatment.
Immune-TACE PFS | 1 year
  Immune-TACE PFS: defined as the time from the first TACE or atezolizumab bevacizumab (whichever occurs first) to the occurrence of one of the following events (whichever occurs first):
  * 20% enlargement of intra- or extra-hepatic lesions as assessed by mRECIST or appearance of new extra-hepatic lesions;
  * TACE refractoriness: insufficient tumor response in the treated tumor for three consecutive times (20% increase by mRECIST);
  * Deterioration of macrovascular invasion (MVI, defined as tumor invasion of the portal vein or hepatic vein and its branches);
  * Deterioration of liver function to Child-Pugh C or mALBI 2b;
  * Death from any cause.
Disease control rate | 1 year
  Disease control rate (DCR): defined as the proportion of patients achieving complete response (CR) or partial response (PR) or stable disease (SD).
Treatment pattern | 1 year
  Treatment pattern: including the timing and frequency of TACE (including its matching chemotherapy regimen), the treatment regimen of atezolizumab + bevacizumab, the sequence of combination therapy and the treatment regimen of the latter line.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital

IPD SHARING:
Plan to Share IPD: Undecided